CLINICAL TRIAL: NCT00439530
Title: Pharmacologic Study of Oseltamivir in Healthy Volunteers
Acronym: SEA002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Southeast Asia Influenza Clinical Research Network (Unknown)
Responsible Party: Yupaporn Wattanagoon, Faculty of Tropical Medicine, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: SEA Trial 0002; SEA ICRN
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2006-11

CONDITIONS: Avian Influenza A Virus
Keywords: oseltamivir; pharmacokinetics; probenecid; avian influenza
MeSH Terms: conditions — Influenza in Birds | interventions — Oseltamivir; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: oseltamivir
Drug: probenecid

SUMMARY:
"Pharmacologic Study of Oseltamivir in Healthy Volunteers" is a Phase I study in which 8 to 32 adult healthy Thai volunteers will be randomized to one of four drug doses and regimens within each of 4 visits. The study is being conducted at the Bangkok Hospital of Tropical Diseases Research Unit, Faculty of Tropical Medicine, and commenced enrolling healthy volunteers on 23 November 2006. The duration of the study is expected to be approximately four months. The goals of this study are to assess the use of loading dose oseltamivir and the concomitant use of probenecid and to characterize the pharmacokinetic properties of oseltamivir in Thai subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy with no underlying chronic disease
* normal baseline laboratory screening
* no regular prescribed medication used in the past 30 days and no over-the-counter medication in the past week
* agree to abstain from self-medication during the study
* negative urine pregnancy test for females and agreement that they will not try to become pregnant until 1 month after the study is completed
* only use non-hormonal methods of contraception for females
* non-smoker for the last 30 days and for duration of the study
* no consumption of alcohol for the last 30 days and for duration of the study
* no use of recreational drugs for the last 30 days and for duration of the study

Exclusion Criteria:

* known hypersensitivity to oseltamivir and/or probenecid
* Hepatitis B virus surface antigen positive
* presence of intercurrent illness or any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
AUC 0-12 hrs. | 12 hour

SECONDARY OUTCOMES:
AUC 12-24 hrs. | 24 hrs
C max | 24 hrs
t max | 24 hrs
t 1/2 | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Yupaporn Wattanagoon, DTM & H, Principal Investigator — Associate Professor, Department of Clinical Tropical Medicine Faculty of Tropical Medicine, Mahidol University
Locations (1):
- Bangkok Hospital for Tropical Diseases Research Unit, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand